CLINICAL TRIAL: NCT00393159
Title: The Influence of The Ear Popper on Serous Otitis Media and on the Accompanying Conductive Hearing Loss in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC06YO3567CTIL
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Otitis Media; Conductive Hearing Loss
Keywords: Effusion; Otitis; Media; Ear; Popper; Children
MeSH Terms: conditions — Otitis Media; Hearing Loss, Conductive; Otitis

INTERVENTIONS:
Device: Ear Popper

SUMMARY:
This study is designed to check the effect of the use of the ear popper device on serous otitis media in children and on the conductive hearing loss accompanying the otitis. It is intended that 30 children aged 3-18 years will participate in the study. The inclusion criteria are : clinical serous otitis media for a duration of more then 3 months, a conductive hearing loss of at least 15 decibels air bone gap and tympanometry type B or C. The children will use the ear popper for 7 weeks. They will undergo otologic examination, audiometry and tympanometry at the beginning ao the trial, at 7 weeks and at 3 months from the beginning of the trial. The otologic findings and the audiometry and tympanometry results before and after the trial will be compared. We will try to determine whether the use of the ear popper in the test group will improve the conductive hearing loss and prevent the need for tympanostomy tube insertion.

ELIGIBILITY:
Inclusion Criteria:

* Serous Otitis Media for More Then 3 months
* Conductive Hearing Loss of More Then 15 decibels.
* Tympanometry type B or C.

Exclusion Criteria:

* No History of Tympanostomy Tube Insertion or Adenoidectomy
* No Cranio or Facial Malformations
* No Acute Upper Respiratory Tract Infection or Acute Otitis Media

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2006-10

PRIMARY OUTCOMES:
Audiometry and tympanometry test results at at 7 weeks and 3 months from beginning of use of the ear popper.
Otoscopic findings at at 7 weeks and 3 months from beginning of use of the ear popper.

SECONDARY OUTCOMES:
Hearing improvement at 7 weeks and 3 months from the beginning of the trial.
Rate of referrals for tympanostomy tube insertion at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yael Oestreicher, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- ENT Unit, Dana Children's Hospital, Tel-Aviv Medical Center, Tel Aviv, Israel